CLINICAL TRIAL: NCT00080912
Title: A Phase III International Randomized Trial Of Single Versus Multiple Fractions For Re-Irradiation Of Painful Bone Metastases
Brief Title: Single vs Multiple-Fraction Therapy in Treating Patients With Previously Irradiated Painful Bone Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network); Trans Tasman Radiation Oncology Group (Other); Cancer Research UK (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC20; CAN-NCIC-SC20 (Other: PDQ); RTOG-0433 (Other: RTOG); TROG-03.08 (Other: TROG); CDR0000357423 (Other: PDQ); NCT00797173 (obsolete NCT alias)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Cancer; Pain
Keywords: bone metastases; pain
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive single-fraction radiotherapy (8 Gy) on day 1.
  Interventions: Radiation: radiation therapy
- Arm II (Active Comparator): Patients receive multiple-fraction radiotherapy (to a total of 20 Gy) over 5 days or over 8 days if re-irradiation of the spine and/or whole pelvis is involved AND prior initial radiotherapy was given in multiple fractions.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Given in a single fraction or multiple fractions

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether single-fraction (single-dose) re-irradiation therapy is as effective as multiple-fraction (many small doses of radiation therapy) re-irradiation therapy in relieving bone pain caused by bone metastases.

PURPOSE: This randomized phase III trial is studying single-dose radiation therapy to see if it works as well as multiple-dose radiation therapy in treating patients previously irradiated with painful bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare pain relief in patients undergoing single-fraction vs multiple-fraction re-irradiation of painful bone metastases at 2 months after treatment.

Secondary

* Compare overall pain relief in patients treated with these regimens.
* Compare time to pain progression in patients treated with these regimens.
* Assess relationship between response to initial radiation and pain relief after re-irradiation in these patients.
* Compare changes in functional interference after re-irradiation using the Brief Pain Inventory in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens (patients in Canada, France, the Netherlands, and patients registered through RTOG).
* Determine characteristics of non-responders (to both initial and re-irradiation) among patients treated with these regimens.
* Monitor the incidence of acute severe radiation-related side effects in patients treated with these regimens.
* Monitor the incidence of in-field pathological fractures and spinal cord compression in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to response to initial radiotherapy (yes vs no), initial fractionation (single fraction vs multiple fraction), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive single-fraction radiotherapy (8Gy) on day 1.
* Arm II: Patients receive multiple-fraction radiotherapy (to a total of 20Gy) over 5 days or over 8 days if re-irradiation of the spine and/or whole pelvis is involved AND prior initial radiotherapy was given in multiple fractions.

At least 4 weeks after the first re-treatment, patients in both arms may receive a second re-treatment at the discretion of the treating oncologist.

Patients complete a Brief Pain Inventory questionnaire at baseline, on days 7 and 14, monthly during months 1-6, and at months 9 and 12. Acute Toxicities are assessed on days 7 and 14. Quality of Life is assessed at baseline and then monthly during months 1-6 for patients from participating groups.

Patients are followed for up to 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 850 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy

  * Diagnosis by needle biopsy, bone marrow biopsy, cytology, or surgical biopsy or resection
* Bone metastases at clinically painful areas confirmed by any of the following:

  * Plain radiographs
  * Radionuclide bone scans
  * CT scans
  * Magnetic resonance imaging
* Worst pain score of ≥ 2/10 using the baseline Brief Pain Inventory
* Pain arising from previously irradiated metastases and not from progressive disease in adjoining or remote areas
* Initial radiotherapy field is reproducible for re-irradiation

  * Current treatment field for palliative radiotherapy must be the same size or smaller than the initial treatment field
* No clinical or radiological evidence of pathological fractures in the target site extremities.
* No radiological evidence of high-risk lesions for pathological fractures in the extremities (lytic lesions > 3cm or > 50% cortical erosion of bone diameter) if target site AND patient is a candidate for surgical intervention.
* No clinical or radiological evidence of spinal cord compression at target site.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective barrier contraception
* Able and willing to complete quality of life questionnaire in English, French, Dutch, or Spanish (if randomized by Canadian, Dutch, French or RTOG centre)
* Must be accessible for treatment follow-up
* Informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No more than 1 prior course of radiotherapy to the target site
* No prior radiotherapy dose ≥ 24 Gy in 6 fractions, 27 Gy in 8 fractions, or 30 Gy in 10 fractions to the spine or any part of the pelvis encompassing small or large bowel and/or the rectum, if these sites are being treated on study

  * Initial doses of 24 Gy in 6 fractions, 27 Gy in 8 fractions or 30 Gy in 10 fractions to the acetabulum or hip and proximal femur allowed as long as the medial field border of the initial treatment did not cross midline
* No prior radiotherapy dose > 30Gy in 10 fractions to the ribs or extremities if these sites are being treated on study
* More than 30 days since prior strontium chloride Sr 89
* More than 30 days since prior half-body radiotherapy, including the current re-irradiation field
* At least 4 weeks since initial radiotherapy

Surgery

* No prior palliative surgery in treatment area
* No concurrent surgical intervention on treatment area

Other

* No prior participation on this protocol
* No plan to make an immediate change in analgesic regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2004-01-22 (Actual); Primary Completion 2013-04-10 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; William F. Hartsell, MD, Study Chair — Advocate Good Samaratin Cancer Centre; Daniel Roos, MD, Study Chair — Royal Adelaide Hospital Cancer Centre; Yvette von der Linden, Study Chair — Radiotherapeutic Institution Friesland; Peter Hoskin, Study Chair — Mount Vernon Cancer Centre
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow E, Hoskin PJ, Wu J, Roos D, van der Linden Y, Hartsell W, Vieth R, Wilson C, Pater J. A phase III international randomised trial comparing single with multiple fractions for re-irradiation of painful bone metastases: National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) SC 20. Clin Oncol (R Coll Radiol). 2006 Mar;18(2):125-8. doi: 10.1016/j.clon.2005.11.014. No abstract available. PMID 16523812
- [Result] Chow E, van der Linden YM, Roos D, Hartsell WF, Hoskin P, Wu JS, Brundage MD, Nabid A, Tissing-Tan CJ, Oei B, Babington S, Demas WF, Wilson CF, Meyer RM, Chen BE, Wong RK. Single versus multiple fractions of repeat radiation for painful bone metastases: a randomised, controlled, non-inferiority trial. Lancet Oncol. 2014 Feb;15(2):164-71. doi: 10.1016/S1470-2045(13)70556-4. Epub 2013 Dec 23. PMID 24369114
- [Derived] Chow R, Ding K, Ganesh V, Meyer RM, van der Linden YM, Roos D, Hartsell WF, Hoskin P, Wu JSY, Nabid A, van Acht M, Wanders R, Babington S, Demas WF, Wilson CF, Wong RKS, Brundage M, Zhu L, Chow E. Gender and age make no difference in the re-irradiation of painful bone metastases: A secondary analysis of the NCIC CTG SC.20 randomized trial. Radiother Oncol. 2018 Mar;126(3):541-546. doi: 10.1016/j.radonc.2017.10.006. Epub 2017 Nov 5. PMID 29102263
- [Derived] Chow E, Meyer RM, Chen BE, van der Linden YM, Roos D, Hartsell WF, Hoskin P, Wu JS, Nabid A, Tissing-Tan CJ, Oei B, Babington S, Demas WF, Wilson CF, Wong RK, Brundage M. Impact of reirradiation of painful osseous metastases on quality of life and function: a secondary analysis of the NCIC CTG SC.20 randomized trial. J Clin Oncol. 2014 Dec 1;32(34):3867-73. doi: 10.1200/JCO.2014.57.6264. Epub 2014 Oct 27. PMID 25349296

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-fraction: Patients receive single-fraction radiotherapy (8 Gy) on day 1.
  radiation therapy: Given in a single fraction or multiple fractions
- Multiple-fraction: Patients receive multiple-fraction radiotherapy (to a total of 20 Gy) over 5 days or over 8 days if re-irradiation of the spine and/or whole pelvis is involved AND prior initial radiotherapy was given in multiple fractions.
  radiation therapy: Given in a single fraction or multiple fractions
Period: Overall Study
Arm/Group | Single-fraction | Multiple-fraction
Started | 425 | 425
Completed | 425 | 425
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-fraction | Multiple-fraction | Total
Number analyzed (Participants) | 425 | 425 | 850
Age, Continuous [Median (Full Range); unit: years] | 64.6 [18.4 to 94.5] | 65.3 [32.0 to 93.0] | 65.1 [18.4 to 94.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient in the single-fraction arm and two patients in the multiple fractions arm have missing sex information.
  Participants
    number analyzed (Participants) | 424 | 423 | 847
    Female | 181 | 167 | 348
    Male | 243 | 256 | 499

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief Measured by the Brief Pain Inventory at 2 Months After Treatment
Description: The primary endpoint of this study is Overall Response Rate (complete response and partial response) at two months after the first fraction of re-irradiation. A complete response was defined as a Brief Pain Inventory worst-pain score of zero with no associated increase in daily oral morphine equivalent. A partial response was defined as pain that persisted after treatment, either with a worst-pain score reduction of 2 or more and no increase in daily oral morphine equivalent consumption, or no increase in pain and a reduction in daily oral morphine equivalent consumption of at least 25%.
Time Frame: 2 months
Population: Intend to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction | Multiple-fraction
Number analyzed (Participants) | 425 | 425
percentage of participants | 28.0 [24.0 to 32.0] | 32.0 [27.0 to 36.0]
Statistical Analysis 1: Comparison: Single-fraction vs Multiple-fraction; Test type: Non-Inferiority or Equivalence — The original sample size was determined based on the non-inferiority. The original sample size is based on assumption of response rate on the multiple fraction arm is 70%, 260 patients were required in each treatment arm to have 80% power to exclude, with a one sided alpha of 0.05, a response rate of 60% or less in the single fraction radiation group (non-inferiority margin =10%). Given an inevaluability rate of 30%, 850 patients (425 for each treatment arm) were randomized to the study; p = 0.03, Cochran-Mantel-Haenszel — p-value is for one-sided non-inferiority test; Risk Difference (RD) = 4.0, 95% CI 1-sided [upper limit 9.2] — The upper limit of one-sided 95% CI for the response rate difference was 9.2%, which was below the pre-specified 10% non-inferiority boundary

ADVERSE EVENTS:
Time Frame: 8.2 years
Arm/Group | Single-fraction | Multiple-fraction
All-Cause Mortality (participants affected / at risk) | 227/425 | 220/425
Serious Adverse Events (participants affected / at risk) | 1/425 | 0/425
Other Adverse Events (participants affected / at risk) | 0/425 | 0/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-fraction (N=425) | Multiple-fraction (N=425)
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No